CLINICAL TRIAL: NCT01957059
Title: A Phase I/II, Open-label, Dose Escalating With 48 Week Treatment Study to Assess the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of BMN053 (Previously Known as PRO053) in Subjects With Duchenne Muscular Dystrophy.
Brief Title: A Phase I/II Study of BMN053 in Subjects With Duchenne Muscular Dystrophy (DMD)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO053-CLIN-01
Record Dates: First submitted 2013-07-02; First posted 2013-10-08 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Duchenne muscular dystrophy; Duchenne; BMN053; BioMarin
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose escalation phase (Experimental): In the dose-escalation phase, following screening assessment, two cohorts of three subjects each receive two single doses of BMN 053 in two study periods (i.e., four single doses in total per subject). In each study period they will receive BMN 053 by IV infusion and by SC injection (separated by one week). The proposed doses are 1 mg/kg (Cohort 1, study period 1), 3 mg/kg (Cohort 2, study period 1), 6 mg/kg (Cohort 1, study period 2) and 9 mg/kg (Cohort 2, study period 2). The actual doses may be amended or repeated based on emerging data from previous doses.
  Interventions: Drug: Regimen Selection Phase Group 1 (COMPLETED)
- Regimen selection (Experimental): After completion of the dose-escalation period of Cohort 1, the safety data of the subjects will be reviewed by a DSMB and if no safety concerns these subjects will continue to receive 6 mg/kg BMN053 weekly by SC injection for 48 weeks. 3 more treatment-naïve subjects will be entered into this Group. These 6 subjects will form Group 1 of the Regimen Selection phase who received 6 mg/kg SC. At the time of this amendment (4) this part of the study has been completed. Following completion of the dose-escalation study period of Cohort 2 (9 mg/kg), the planned review of the preliminary plasma PK data from the dose-escalation phase showed a relative bioavailability of 50% for BMN053 with SC dosing (50% lower plasma AUC after SC dosing compared to IV dosing). Taking into consideration the risk of injection site reactions noted with similar compounds when administered SC over longer term, the planned 9 mg/kg BMN053 weekly by SC injection will be discontinued to be replaced by an IV regimen.
  Interventions: Drug: Regimen Selection Phase Group 2; Drug: Regimen Selection Phase Group 3
- 48-week Treatment Phase (Experimental): Thirty additional treatment-naïve subjects will be recruited for the primary evaluation and will receive treatment at the recommended regimen for a total of 48 weeks. Subjects dosed initially in the dose escalation phase and/or the regimen selection phase of the study will not be included in the primary analysis.
  Following completion of the 2nd study period for Cohort 2, the safety data will be reviewed by the DSMB and in the absence of safety concerns the subjects may enter the 48 week treatment phase and receive 9 mg/kg PRO053 once weekly by SC injection. Three new subjects will enter cohort 2 (i.e. 6 subjects in total at this dose level).
  After the initial 12 subjects have completed 12 weeks of dosing the dose for the Treatment group (30 new subjects) will be selected based on the totality of the 12-week data from those initial 12 subjects. The initial 12 subjects will also be dosed on the selected dose (i.e. continue on their dose or [down-]titrate).
  Interventions: Drug: Treatment Phase Group 4
- Dosing extension (Experimental): All subjects who have completed the dose escalation and regimen selection phase of the study (N=15), and subjects who have complete the treatment phase of the study who have tolerated the treatment will be offered to continue dosing in the dosing extension with ongoing assessment of efficacy, safety, and tolerability of BMN 053. Safety, efficacy, PK/PD and biomarker assessments will be performed at scheduled visits; adverse events (AEs) and concomitant medications and therapies will be continuously monitored. The dose extension phase will provide BMN 053 treatment for 48 weeks.
  Interventions: Drug: Dosing Extension

INTERVENTIONS:
Drug: Regimen Selection Phase Group 2 — All doses of BMN053 will be administered as IV infusions. The proposed doses are as follows:
  • 3 mg/kg
  Arms: Regimen selection
Drug: Regimen Selection Phase Group 3 — All doses of BMN053 will be administered as IV infusions. The proposed doses are as follows:
  • 4-6 mg/kg
  Arms: Regimen selection
Drug: Treatment Phase Group 4 — All doses of PRO053 will be administered as IV infusions. The proposed doses will be decided upon completion of the Regimen Selection Phase of Groups 2 and 3
  Arms: 48-week Treatment Phase
Drug: Regimen Selection Phase Group 1 (COMPLETED) — All doses of BMN053 have been administered as subcutaneous injections.
  Arms: Dose escalation phase
Drug: Dosing Extension — All doses of PRO053 will be administered as IV infusions. The proposed doses will be decided upon completion of the Regimen Selection Phase of Groups 2 and 3 and the Treatment Phase Group 4.
  Arms: Dosing extension

SUMMARY:
The purpose of the study is to see whether BMN053 is safe and effective to use as medication for Duchenne muscular dystrophy (DMD) patients with a mutation around location 53 in the DNA for the dystrophin protein.

DETAILED DESCRIPTION:
A Phase I/II, open-label, dose escalating with 48-week treatment study to assess the safety and tolerability, pharmacokinetics, pharmacodynamics and efficacy of BMN 053 (previously known as PRO053) in subjects with Duchenne muscular dystrophy

ELIGIBILITY:
Inclusion Criteria:

1. Duchenne muscular dystrophy resulting from a mutation correctable by treatment with BMN053 confirmed by a state-of-the-art DNA diagnostic technique covering all DMD gene exons, including but not limited to MLPA (Multiplex Ligation-dependent Probe Amplification), CGH (Comparative Genomic Hybridisation), SCAIP (Single Condition Amplification/Internal Primer) or HRMCA (High-Resolution Melting Curve Analysis).
2. Ambulant boys aged at least 5 years on the day of first dosing able to walk for at least 300 metres in the 6 minute walking distance (6MWD) test. In addition, results of the 6MWD test must be within ±30 metres of each other at 2 of 3 pre-treatment visits (screen 1, 2 and baseline) prior to first BMN053 administration.
3. Adequate quality for biopsy (confirmed with MRI) of the lateral head of the gastrocnemius muscle. Only under exceptional circumstances will an alternative muscle (preferably brachii) be considered for biopsy and only following discussion between the Principal Investigator and the BioMarin Medical Monitor.
4. Life expectancy of at least 3 years after inclusion in the study.
5. Glucocorticosteroid use which is stable for at least 3 months prior to first BMN053 administration. Subjects must have been receiving glucocorticosteroids for at least 6 months prior to the first BMN053 administration.
6. Willing and able to adhere to the study visit schedule and other protocol requirements.
7. Written informed consent signed (by parent(s)/legal guardian and/or the subject, according to the local regulations).
8. In France, a subject will be eligible for inclusion in this study only if either affiliated to, or a beneficiary of, a social security category.
9. Anticipated adequate vein access for intravenous (IV) infusion.

Exclusion Criteria:

1. Current or history of liver disease or impairment.
2. Current or history of renal disease or impairment.
3. At least two aPTT above upper limit of normal (ULN) within the last month prior to first dose of BMN053.
4. Screening platelet count below the lower limit of normal (LLN).
5. Acute illness within 4 weeks prior to first dose of BMN053 which may interfere with the study assessments.
6. Severe mental retardation and/or behavioural problems which, in the opinion of the Investigator, prohibit participation in this study.
7. Severe cardiomyopathy which, in the opinion of the Investigator prohibits participation in this study. If a subject has a left ventricular ejection fraction <45% at screening, the Investigator should discuss inclusion of the subject with the Medical Monitor.
8. Expected need for daytime mechanical ventilation within the next year.
9. Use of anticoagulants, antithrombotics or antiplatelet agents.
10. Use of idebenone or other forms of coenzyme Q10 within 1 month prior to the start of the screening for the study.
11. Use of nutritional or herbal supplements which, in the opinion of the Investigator, may influence muscle performance within 1 month prior to first dose of BMN053.
12. Use of any other investigational product or participation in another trial with an investigational product, within 6 months prior to the start of the screening for the study.

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-08-03 (Actual); Study Completion 2016-08-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 6 minute walk test | after 48 weeks of treatment phase

SECONDARY OUTCOMES:
Muscle function | after 48 weeks treatment phase
Muscle strength | after 48 weeks treatment phase
Pulmonary function | after 48 weeks treatment phase
Functional outcomes questionnaire | after 48 weeks treatment phase
Adverse Events | after single intravenous and subcutaneous doses, and after 48 weeks of treatment phase
Safety Laboratory | after single intravenous and subcutaneous doses, and after 48 weeks of treatment phase
Cardiac function | after single intravenous and subcutaneous doses, and after 48 weeks of treatment phase
Pharmacokinetic parameters at different dose levels | after single intravenous and subcutaneous doses, and after 48 weeks of treatment phase
Presence of (BMD-like) dystrophin expression in muscle biopsy | after 48 weeks treatment phase
Production of exon skip 53 mRNA in muscle biopsy | after 48 weeks treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: V. Straub, Prof., Principal Investigator — Institute of Genetic Medicine, Newcastle University, UK
Locations (6):
- UZ Leuven, Campus Gasthuisberg, Leuven, Belgium
- Institut de Myologie, Paris, France
- Policlinico Universitario Agostino Gemelli, Rome, Italy
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- United Kingdom (2):
  - Great Ormond Street Hospital for Children, London
  - Institute of Genetic Medicine International Centre for Life, Newcastle

REFERENCES:
- See also: BioMarin website — http://www.biomarin.com